CLINICAL TRIAL: NCT02735785
Title: Adapting the HOPE Social Media Intervention to Reduce Prescription Drug Abuse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sean Young, PhD, MS, Assistant Professor of Family Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21DA039458 (NIH)
Record Dates: First submitted 2016-02-05; First posted 2016-04-13 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Non-Cancer Chronic Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- intervention (Experimental): behavioral intervention
  Interventions: Behavioral: Harnessing Online Peer Education (HOPE) Social Media Intervention
- control (No Intervention): control

INTERVENTIONS:
Behavioral: Harnessing Online Peer Education (HOPE) Social Media Intervention
  Arms: intervention

SUMMARY:
The Harnessing Online Peer Education (HOPE) intervention combines social media with a psychology-based interventions to change behavior. This intervention is being applied to reduce prescription drug abuse among patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* (a) UCLA health system patient,
* (b) ≥ 18 years of age,
* (c) on chronic opioid therapy (> 3 and < 12 months) for chronic non-cancer pain as reported by their physician who referred them.

Exclusion Criteria:

° Does not satisfy inclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Current Opioid Misuse Measure (COMM) Score | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States